CLINICAL TRIAL: NCT02347319
Title: A Double-Blind, Randomized, Multicenter Trial Examining the Efficacy of Biphenyl Dimethyl Dicarboxylate Combined With Garlic Oil in Patients With Transaminase Elevated Chronic Liver Disease
Brief Title: To Evaluate the Efficacy of DDB/Garlic Oil in Patients With Elevated Transaminase Chronic Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P2010-PN004
Record Dates: First submitted 2013-06-11; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Liver Disease
MeSH Terms: interventions — Silymarin; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pennel (Experimental): This group will treated with DDB 25mg/Garlic oil 50mg for 12 weeks.
  Interventions: Drug: Pennel
- Legalon (Active Comparator): This group will treated with Silymarin 140mg for 12 weeks.
  Interventions: Drug: Legalon
- Placebo (Placebo Comparator): This group will treated with Placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pennel — Pennel 2 Tablet, Legalon Placebo 1 tablet, Tid
  Other Names: DDB/Garlic oil
  Arms: Pennel
Drug: Legalon — Pennel Placebo 2 Tablet, Legalon 1 tablet, Tid
  Other Names: Silymarin
  Arms: Legalon
Drug: Placebo — Pennel Placebo 2 Tablet, Legalon Placebo 1 tablet, Tid
  Other Names: Lactose
  Arms: Placebo

SUMMARY:
Purpose

- To evaluate the efficacy of Biphenyl dimethyl dicarboxylate(DDB)/Garlic Oil in patients with elevated transaminase chronic liver disease.

DETAILED DESCRIPTION:
Biphenyl dimethyl dicarboxylate (DDB) combined with garlic oil (pennel) has been used to treat chronic liver disease. A randomized, double-blind, active- and placebo-controlled clinical trial was conducted to investigate the efficacy, safety and quality of life in chronic liver disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 20years of age
* Patients with more 60 ALT in screening period.
* To evaluate ALT and AST at least three months.
* Serum Transaminase abnormal(before 6months), chronic liver disease or fatty liver, liver disease medical treatment at more than 30days
* Women of childbearing age get her consent for contraception, pregnancy urine test result negative.

Exclusion Criteria:

* ALT>10UNL on screening period.
* Current treatment on another clinical trial
* Pregnancy or breastfeeding

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Normalized rate in serum ALT | 12 weeks
  The rate of alanine aminotransferase (ALT) normalization

SECONDARY OUTCOMES:
ALT | 8, 12 weeks
AST | 8, 12 weeks
γ-GTP | 8, 12 weeks
AST/ALT ratio | 8, 12 weeks
ALP | 8, 12 weeks
Albumin | 8, 12 weeks
Total Bilirubin | 8, 12 weeks
The assessment of health-related quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The catholic university of korea, Bucheon ST. Mary's Hosipital, Bucheon-si, Gyeonggi-do, South Korea